CLINICAL TRIAL: NCT02897323
Title: Northwest Inter Hospital Adult Congenital Heart Disease Observatory
Brief Title: Northwest Adult Congenital Heart Disease Observatory
Acronym: CARL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 14-140
Record Dates: First submitted 2016-08-29; First posted 2016-09-13 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: description

SUMMARY:
The incidence of congenital heart disease is about 8 per thousand live births. Thanks to advances in cardiac surgery, 90% of children born with heart defects reach adolescence and adulthood. Congenital heart defects are the leading cause of heart disease in young adults and expectant mothers in Western countries. The number of patients increases continuously as life expectancy increases. An increasing number of patients with complex heart defects survive to adulthood. The medico-surgical management of this highly specialized growing number of patients is difficult and requires a multidisciplinary collaboration. In France, an estimated 200,000 patients the number of carrier patients with congenital heart disease. Half of them will require monitoring, medical procedures, catheterizations and/or surgical re-intervention. No objective demographic data are currently available on the French patients. So, the investigators decided to set up an epidemiological project to better understand this cohort of patients. The main objective of this project is to obtain accurate epidemiological data needed to adapt the supply of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 years
* Congenital heart disease operated or non-operated
* Followed by a cardiologist specializing in congenital heart disease in the inter northwest region of France

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients visiting the participating centers meet the following criteria:
  * Patient, male or female, aged 18 years
  * with congenital heart disease operated or non-operated
  * Followed by a cardiologist specializing in congenital heart disease in the inter northwest region of France
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
patients characteristics description | baseline
  Obtain epidemiological data on adult congenital of the population followed in northwest region of France

SECONDARY OUTCOMES:
heart disease complications description | baseline
complications during pregnancy description | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided